CLINICAL TRIAL: NCT07036640
Title: The Impact of Acute Exercise in the Heat on Breast Milk Production and Composition in Lactating Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Providence College (Other)
Responsible Party: Principal Investigator, Margaret Morrissey, Assistant Professor, Providence College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB-FY25-26
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lactation
Keywords: Lactation; Exercise; Heat Stress
MeSH Terms: conditions — Breast Feeding; Motor Activity; Heat Stress Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat exposure (Experimental): Heat exposure in environmental chamber during exercise (60 mins)
  Interventions: Other: Heat exposure
- Thermoneutral Condition (No Intervention): Thermoneutral temperature (non-heat exposure condition)

INTERVENTIONS:
Other: Heat exposure — Heat exposure during exercise
  Arms: Heat exposure

SUMMARY:
This clinical trial aims to determine whether heat stress alters 24-hour breast milk production and composition following an acute bout of exercise in the heat among lactating women.

The main questions are:

1. To ascertain whether heat stress alters 24-hour breast milk production following acute exercise in the heat among lactating women. We hypothesize that breast milk production will decrease to a greater extent following acute exercise in the heat compared to acute exercise with no heat stress. Lactating mothers will complete an acute exercise bout at 40% of their peak oxygen consumption (VO2peak) for 60 mins in a hot (36 °C, 40% relative humidity) and thermoneutral environment (20 °C, 20% relative humidity). Participants will record their total breast milk production in a 24-hour period using an infant scale.
2. to discover whether heat stress impacts the energy composition of breast milk following acute exercise in the heat among lactating women. We hypothesize that energy density will decrease to a greater extent following acute exercise in the heat compared to acute exercise with no heat stress. Participants will use a manual expression breast pump to collect 10 mL of breast milk from each breast immediately and 24 hours post-exercise. Energy density (lactose, protein, and lipid content) will be assessed via enzyme-linked immunosorbent assays.

Participants will complete the following visits: 1) initial consent visit 2) baseline testing; 3) acute exercise in the hot condition (HOT; 36C, 40% relative humidity), and 4) acute exercise in the temperate, thermoneutral condition (TEMP; 20C, 20% relative humidity). The baseline testing day will measure participant anthropometrics including height, weight, and body composition measured by a DEXA scan. For both experimental trials, participants will be asked to walk on a treadmill at based on their metabolic heat production (8W/kg) for 60 minutes. Heart rate (HR), mean skin temperature (Tsk), core temperature (Tcore), sweat loss (SL), and fluid intake will be measured throughout the exercise protocol. Breast milk composition will be measured through milk expression using a manual expression breast pump immediately and 24 hours post-exercise. Participants will log their breast milk production for 24 hours following the exercise using an infant scale to measure their infants before and after each feed.

DETAILED DESCRIPTION:
This study will be a randomized, cross-over design with four study visits: 1) an initial visit where the participant can see the study equipment, ask questions, and fill out a brief questionnaire to determine whether they are eligible to participant; 2) baseline and metabolic heat production testing; 3) acute exercise in the hot condition [experimental trial 1 (HOT): 36C, 40% relative humidity], and 4) acute exercise in the temperate, thermoneutral condition [experimental trial 2 (TEMP): 20C, 20% relative humidity]. Data collection will occur at the Health and Human Performance Laboratory (HHPL) in the Department of Health Sciences.

Visit 1: Initial Visit The participant will come to the lab for an initial visit. During this brief visit (<30 min), the participant can ask questions about the study, see the study equipment, and will be asked to complete a questionnaire to determine their eligibility.

Visit 2 (Baseline and Metabolic Heat Production Testing):

The baseline testing will collect participant anthropometric data, which includes height, body mass, and body composition (dual-energy X-ray absorptiometry, DXA) scan and a stepwise metabolic heat production test. Participants will report to the laboratory having abstained from caffeine, alcohol, and food (12, 24, and 4 hours, respectively). Upon arrival, participants will provide a small urine sample in a sterile urine cup to measure hydration status and for a pregnancy test. Researchers will measure hydration status using a refractometer. If the pregnancy test is positive, the PI will inform the participant that the test is positive and will not perform the scan. The participant will also no longer be eligible to continue with the study. After hydration assessment, nude body mass and height will be collected and the participant's body composition will measured using DXA. To obtain a nude body mass, a private curtain-changing area with a body weight scale will be provided to ensure privacy. Only the participant will be able to enter. The scale reading will come outside the private curtain area for the researchers to see. The DXA software will generate lean mass, fat mass, and body fat percentage. To calculate exercise intensity based on a fixed metabolic heat production (per unit body mass), participants will undergo a 24-min incremental treadmill test in an environmental chamber. Participants will perform the test in the same environmental conditions as the HOT trial (36C, 40% relative humidity; described below). Participants will don a heart rate (HR) monitor before testing. The treadmill test will consist of 6 x 4-min stages and progressively increase speed (2.5mph, 3.0mph, 3.5mph, 4.0mph, 4.5mph, and 5.0mph). The treadmill grade will be set at 2% to account for terrain and wind resistance. Oxygen consumption and respiratory exchange were collected continuously (30-sec average) using a Hans Rudolph metabolic mask (Hans Rudolph Inc., Shawnee, KS, USA) attached to a hose and delivered to the metabolic cart system (Parvo Medics Truemax 2400 Metabolic Measurement System, Consentius Technologies, Sandy, UT). These variables will be used to calculate metabolic heat production using partitional calorimetry (Cramer & Jay, 2019). An exercise intensity of 8 W/kg was selected to elicit a brisk walking intensity. The metabolic heat production test is a standard procedure used in the thermal physiology literature to perform an unbiased comparison of thermoregulatory responses between groups (Jay & Cramer 2015).

Visit 3 and 4: Experimental Trials (HOT & TEMP). Experimental trials (HOT and TEMP) will consist of a 60 min treadmill exercise protocol at a fixed metabolic heat production per unit body mass (8 W/kg). Exercise will be performed in an environmental chamber. HR, mean skin temperature (Tsk), core temperature (Tcore), sweat loss, and fluid intake will be measured throughout the exercise protocol. Breast milk composition will be measured through milk expression using a manual expression breast pump 24-hour before (post exercise), one hour-post exercise and 24 hours post-exercise. Breastmilk samples will not be collected at the laboratory. Participants will be asked to collect samples at home and will be provided written instructions on the breastmilk collection procedure (described below). Participants will log their breast milk production for 24 hours before and after the exercise protocol using a supplied infant scale.

Over 24 hr before the start of exercise, participants will be provided with a water bottle to track their fluid intake, Tcore pill, food log, an infant scale, breastmilk production log, manual breastmilk expression pump, storage bag, and small cooler bag for transport. Participants will log their food and fluid intake during the day before, during, and after each experimental trial (24 hr before and after). Participants will be asked to maintain similar dietary habits during either experimental session. Participants will also be given an ingestible pill thermistor for Tcore assessment and asked to consume one pill approximately 6 hours before the start of exercise. Twenty-four hours before the start of the trial, participants will be asked to manually express 5 mL of breast milk immediately before the infant is put on the breast and 5 mL immediately after the infant has finished suckling. Participants who only express breastmilk will collect 5 mL from the start and end of their breastmilk expression session. This will collect fore and hind breast milk samples to account for different lipid concentrations between milk types. The fore and hind breastmilk samples will be analyzed separately and entered into a formula to estimate energy density [2,3] Breastmilk samples will be stored in the breastmilk storage bag provided. Participants will be asked to store the breast milk in their refrigerator and use the provided cooler bag to transport breastmilk when arriving for their visit. Participants will be asked to log breastmilk production by weighing infants (test weighing) or the quantity of expressed breast milk (see weighing infant protocol below).

On the experimental trial days, participants will report to the laboratory in the morning. Hydration status will be assessed through urine-specific gravity, urine color assessment, and body mass changes. If the core temperature pill passes before visit, the participant will have the option to use a core temperature pill as a suppository or re-schedule their trial. The pill will be given to you at your initial visit. Participants will be asked to wear an HR monitor and four skin temperature sensors placed on their chest, shoulder, thigh, and calf to assess mean Tsk. Participants will enter the environmental chamber for the exercise protocol. Immediately upon entering the environmental chamber, participants will perform a seated 10-minute passive equilibration period. Participants will then walk briskly at 8 W/kg for 60 mins. During exercise, Tcore, Tsk, and HR will be continuously monitored. Fluid will not be permitted during exercise.

After completing the exercise protocol, participants will provide a urine sample for hydration assessment, and body mass will be measured. Participants will receive a water bottle to track their fluid intake, food log, an infant scale (Doran DS4500), breastmilk production log, manual breastmilk expression pump, storage bag, and small cooler bag for transport before leaving the laboratory. Participants will be asked to log breastmilk production by weighing infants (test weighing) or the quantity of expressed breast milk. To account for evaporative losses, participants will be asked to measure their infants immediately before (Wb), immediately after (Wa), and 20 min (We) after feeding [4]. One hour and 24 hours after the completion of the exercise, participants will be asked to provide breast milk samples. Participants will be asked to store the breast milk in their refridgerator and use the provided cooler bag to transport breastmilk when arriving for their last visit (Visit 3). Following Visit 3, researchers will ask participants to report to the laboratory with frozen breast milk storage and to return other supplies (i.e., infant scale, manual breastmilk expression pump).

When participants bring in their breastmilk samples, fat content within them will be assessed immediately using the Creamatocrit method (Miller et al. 2013). Three mL of each sample will be aliquoted into separate 1-mL creamatocrit collection tubes. Each 1-mL milk sample will be placed into a micro-capillary tube and centrifuged for 3-5 minutes around 10,000 rpm. The height of the fat layer and total milk column will be measured following centrifugation

The remaining breastmilk sample will be immediately frozen in -80C after collection [5].The protein content of breastmilk samples will be determined using a Pierce Modified Lowry Protein assay kit [5,6] and lactose content will be measured using a lactose colorimetric assay kit after data collection is complete [5,7].

References:

1. Jay O, Cramer MN. A new approach for comparing thermoregulatory responses of subjects with different body sizes. Temperature (Austin). 2015 Feb 11;2(1):42-3. doi: 10.1080/23328940.2014.996093. PMID: 27227002; PMCID: PMC4843865.
2. Miller EM, Aiello MO, Fujita M, Hinde K, Milligan L, Quinn EA. Field and laboratory methods in human milk research. Am J Hum Biol. 2013 Jan-Feb;25(1):1-11. doi: 10.1002/ajhb.22334. Epub 2012 Oct 29. Erratum in: Am J Hum Biol. 2013 May-Jun;25(3):442. PMID: 23109280.
3. Saint L, Smith M, Hartmann PE. 1984. The yield and nutrient content of colostrum and milk of women from giving birth to one month post-partum. BMJ 52:87-95.
4. Woodward DR, Cumming FJ. Do ambient temperature and humidity influence the breast-milk intake of babies? J Paediatr Child Health. 1990;26:347-50. doi: 10.1111/j.1440-1754.1990.tb02450.x
5. Nommsen L, Lovelady C, Heinig M, et al. Determinants of energy, protein, lipid, and lactose concentrations in human milk during the first 12 mo of lactation: the DARLING Study. Am J Clin Nutr. 1991;53:457-65. doi: 10.1093/ajcn/53.2.457
6. PierceTM Modified Lowry Protein Assay Kit. https://www.thermofisher.com/order/catalog/product (accessed 30 July 2024.
7. Lactose Assay Kit (Colorimetric/Fluorometric) | LSBio. https://www.lsbio.com/assaykits/lactose-assay-kit-colorimetric-fluorometric-ls-k289/289 (accessed 30 July 2024)

ELIGIBILITY:
Inclusion Criteria:

* Currently breastfeeding or pumping expressed breastmilk for their 6-week to 24-month infants
* Aged 18-45 years old
* Delivered their infants between 37-42 weeks of gestational age

Exclusion Criteria:

* Obsterical complications during pregnancy
* multiple gestation
* Chronic disease (i.e., diabetes, hypertension, metabolic disease)
* Heat illnness in the last 3 month

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Breastmilk Composition | Measured 24hr before exercise, one hour post-exercise, and 24hr post exercise for each condition
  Breastmilk lipid, protein, and lactose content
Breastmilk Production | Collected 24-hour before exercise, 1-hour post-exercise, and 24-hour post-exercise
  Breastmilk production (lactation)

SECONDARY OUTCOMES:
Core temperature | Collected every minute for 60 minutes during exercise
  Internal core body temperature
Heart rate | Collected every minute for 60 minutes during exercise
  Heart rate
Skin temperature | Collected every minute for 60 min during exercise
  Mean skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Margaret C Morrissey-Basler, PhD, Principal Investigator — Providence College
Locations (1):
- Providence College, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared following the completion of the study.

REFERENCES:
- [Background] Nommsen LA, Lovelady CA, Heinig MJ, Lonnerdal B, Dewey KG. Determinants of energy, protein, lipid, and lactose concentrations in human milk during the first 12 mo of lactation: the DARLING Study. Am J Clin Nutr. 1991 Feb;53(2):457-65. doi: 10.1093/ajcn/53.2.457. PMID 1989413
- [Background] Woodward DR, Cumming FJ. Do ambient temperature and humidity influence the breast-milk intake of babies? J Paediatr Child Health. 1990 Dec;26(6):347-50. doi: 10.1111/j.1440-1754.1990.tb02450.x. PMID 2073422
- [Background] Saint L, Smith M, Hartmann PE. The yield and nutrient content of colostrum and milk of women from giving birth to 1 month post-partum. Br J Nutr. 1984 Jul;52(1):87-95. doi: 10.1079/bjn19840074. PMID 6743645
- [Background] Miller EM, Aiello MO, Fujita M, Hinde K, Milligan L, Quinn EA. Field and laboratory methods in human milk research. Am J Hum Biol. 2013 Jan-Feb;25(1):1-11. doi: 10.1002/ajhb.22334. Epub 2012 Oct 29. PMID 23109280